CLINICAL TRIAL: NCT07150832
Title: I-CARE: Efficacy of a Digital Health Intervention to Reduce Suicidal Ideation During Psychiatric Boarding
Brief Title: Efficacy of the I-CARE Digital Health Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Yale University (Other); Weill Medical College of Cornell University (Other); Dartmouth College (Other)
Responsible Party: Principal Investigator, JoAnna K. Leyenaar, Professor of Pediatrics, Professor of The Dartmouth Institute, Trustees of Dartmouth College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LSRG-1-094-23; STUDY00033318 (Other: Dartmouth College Committee for the Protection of Human Subjects); 2000039368 (Other: Yale Human Research Protection Program Institutional Review Boards); FWA00000093 (Other: Weill Cornell Medicine Research Integrity Institutional Review Board); STUDY02002242 (Other: Dartmouth Health Institutional Review Board)
Record Dates: First submitted 2025-08-28; First posted 2025-09-02 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-08

CONDITIONS: Mental Health Disorder; Suicide Attempt; Suicidal Ideation; Emergency Psychiatric
Keywords: Children; Adolescents; Emergency Department; Mental Health Boarding; Psychosocial Skills
MeSH Terms: conditions — Mental Disorders; Suicide, Attempted; Suicidal Ideation; Emergencies | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-CARE (Experimental): I-CARE (Improving Care, Accelerating Recovery & Education) is a tablet-based program designed to deliver evidence-based psychosocial skills to adolescents during mental health boarding. The program consists of 7 web-based animated videos and workbook exercises, facilitated by non mental health professionals.
  Interventions: Behavioral: Improving Care, Accelerating Recovery & Education (ICARE)
- Safety Supervision (No Intervention): These hospitals currently offer basic safety supervision and medical monitoring for adolescents during mental health boarding. This is the "usual care" condition.

INTERVENTIONS:
Behavioral: Improving Care, Accelerating Recovery & Education (ICARE) — I-CARE is a brief, digital intervention designed for adolescents who are boarding in a medical hospital awaiting transfer to a psychiatric inpatient unit. It consists of 7 tablet-based animated video modules and workbook exercises, facilitated by individuals who are not mental health professionals. All modules are grounded in evidence-based practices, such as cognitive-behavioral therapy and dialectical behavior therapy.
  Arms: I-CARE

SUMMARY:
When presenting to an ED with suicide, self-harm or other mental health crises, youth may also experience "boarding", which is defined by the Joint Commission as "the practice of holding patients in the ED or another temporary location after the decision to admit or transfer has been made." A recent national survey of 88 US acute care hospitals conducted by our research team found that 98.9% of hospitals were boarding youth awaiting psychiatric hospitalization, for an average of 2-3 days. However, as illustrated in a systemic review, little research has focused on developing interventions to support youth during this highly vulnerable time. 3

I-CARE is a modular, blended digital health intervention facilitated by individuals who are not mental health clinical staff to teach youth evidence-based psychosocial skills during the boarding period. This study will evaluate I-CARE's efficacy using a patient-level randomized clinical trial (RCT), randomizing youth to receive standard safety supervision or I-CARE in addition to standard safety supervision. If found to the efficacious, I-CARE could be scaled-up in new settings with limited resources and has the potential to significantly improve the quality of care received by youth experiencing boarding.

DETAILED DESCRIPTION:
Suicide is the second leading cause of death among adolescents; from 2007 to 2017 suicide deaths tripled in youth 10 to 14 years. Emergency departments (EDs) at acute care hospitals increasingly serve as portals of care for youth with suicidal ideation or attempt. When these youth are deemed to require psychiatric hospitalization, the demand for beds often exceeds supply, leading to psychiatric boarding. To address this gap, a multidisciplinary team including pediatricians, psychologists and patient partners developed a modular digital intervention and associated training materials to deliver evidence-based psychosocial skills to youth during boarding. This program, entitled I-CARE (Improving Care, Accelerating Recovery & Education), consists of 7 web-based animated videos and workbook exercises, facilitated by licensed nursing assistants who provide 1-on-1 safety supervision during boarding. Given that 1-on-1 safety supervision is the current standard of care at most hospitals, I-CARE requires minimal additional resources beyond those already available in these settings. The psychosocial skills included in I-CARE are grounded in cognitive behavioral therapy and were prioritized through a rigorous Delphi process evaluating their importance and feasibility to deliver during psychiatric boarding.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents of any sex and gender, aged 12-17 years at ED visit or hospital encounter
* Presenting with suicide attempt or ideation, or self-harm
* Medically stable
* English-speaking
* Awaiting transfer for inpatient psychiatric care or disposition.

Exclusion Criteria:

* Cognitive or developmental delays precluding participation (intellectual functioning <12 years of age)
* Behavioral limitations that preclude program participation
* Active psychosis
* Legal parent/caregiver unable to speak English or unavailable to provide consent (e.g. Wards of the State)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 173 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scales Youth Version (DASS-Y ) | Baseline/hospital admission (T1), hospital discharge/approximately 72 hours after admission (T2), and 30 days (T3), 60 days (T4), and 90 days (T5) post-discharge
  The DASS-Y is a 21-item, youth-oriented validated measure that generates an aggregate assessment of emotional distress and sub-measures of depression, anxiety, and stress. Each item is self-reported on a 4-point Likert scale ranging from 0 (Did not apply to me at all) to 3 (Applied to me very much, or most of the time).
9-item Concise Health Risk Tracking - Self-Report (CHRT-SR9) | Baseline/hospital admission (T1), hospital discharge/approximately 72 hours after admission (T2), and 30 days (T3), 60 days (T4), and 90 days (T5) postdischarge
  The Concise Health Risk Tracking (CHRT) is a 9-item survey that assesses suicidal thoughts and behaviors in the past week, with response options ranging 0-4. Total scores range 0-36, with higher scores indicating more severe suicidality.
Harkavy-Asnis Suicide Scale (HASS) | Time Frame: 30 days (T3), 60 days (T4), and 90 days (T5) postdischarge
  The HASS consists of 21 self-report items that cover the range of suicidal ideation and attempts, including both passive and active ideation. Responses on each item range 0-4; total scores range 0-84, with higher scores indicating more severe suicidality. The study will use only the 2 questions that inquire about suicide attempts.

CONTACTS AND LOCATIONS:
Overall Officials: JoAnna K. Leyenaar, MD, PhD, MPH, Principal Investigator — Dartmouth College
Locations (4):
- United States (4):
  - Yale, New Haven, Connecticut
  - Dartmouth College, Hanover, New Hampshire
  - Dartmouth Health, Lebanon, New Hampshire
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded into the NIMH Data Archive (NDA).
  Data will be collected from approximately 173 adolescents 12-17 years of age. Measures include:
  1. Depression, Anxiety, and Stress Scale - Youth version (DASS-Y)
  2. Harkavy-Asnis Suicide Scale (HASS) - Suicide Attempt module
  3. Concise-Health Risk Tracking-Self Report (CHRT)
  4. Revised Children's Anxiety and Depression Scale-25 (RCADS-25)
Supporting Information: Study Protocol
Time Frame: All data will be deposited to NDA starting 12 months after the award begins and will be deposited every six months thereafter following the usual NDA data submission dates.
Access Criteria: All those with access to the NDA will have access to our data.